CLINICAL TRIAL: NCT01823796
Title: Assessment of Balance and Risk of Falls in Women With Fibromyalgia
Brief Title: Risk of Falls in Patients With Fibromyalgia
Acronym: FM
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assistant professor, Universidad de Granada
Other Study IDs: DF0041G
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; balance; falls
MeSH Terms: conditions — Fibromyalgia | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy women.: 35 healthy women. Control group.
  Interventions: Other: Healthy women
- Fibromyalgia women group: 35 women with fibromyalgia were measured at baseline of the observational study.
  Interventions: Other: Fibromyalgia women group

INTERVENTIONS:
Other: Fibromyalgia women group — Assessment of this group at baseline in order to be compared with a control group.
  Other Names: Fibromyalgia
  Groups: Fibromyalgia women group
Other: Healthy women — These women are assessed in order to be compared with fibromyalgia women group.
  Other Names: Control group
  Groups: Healthy women.

SUMMARY:
Fibromyalgia is a chronic illness characterized by persistent widespread muscle pain with generalised hyperalgesia and allodynia. It can be accompanied by other concomitant symptoms: fatigue, sleep disturbances, musculoskeletal disorders, distress and psychological disorders. The prevalence has been reported to be between 2 and 5%.

The hypothesis of this study is that women with fibromyalgia present high risk of falls and balance disorders compared with healthy women. The objective of this study was to investigate wether gait pattern changes in single and dual task conditions were associated with the risk of falling in women with fibromyalgia.

DETAILED DESCRIPTION:
Falls and fall-related injuries are a common health problem. A fall is often a result of intrinsic physiological ageing and underlying chronic disease interacting with the external and challenging environment. Disturbances in physical function, muscle strength, range of motion, poor balance, affectation in sensory system, a loss of proprioception, alteration concerning visual and vestibular aspects, dizziness, decreased endurance and cognitive and mobility impairment are the most common risk factors for falls. Postural control in a dual task setting is especially relevant to daily life situations. Attending to that, we propose an assessment based on these parameters in women with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with fibromyalgia attending to the Fibromyalgia Association of Granada.
* Women who can complete the assessment battery of tests and tasks.

Exclusion Criteria:

* Auditive and visual disturbances.
* Cognitive problems.
* Psychiatric pathology.
* Gait serious disturbances.
* Concomitant neurological conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with fibromyalgia. Fibromyalgia is a chronic condition characterised by chronic pain, fatigue, sleep disorders and psychological disturbances.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Timed up & Go (TUG) | baseline
  This test timed in seconds measure the time taken by the participant to stand up from an arm chair, walk 3 metres at normal pace, turn around, walk back and sit down. They start to the order of "Go!" A stopwatch was used to measure the time. The TUG is a frequently used test to assess mobility and fall risks in older adults and is recommended by American Geriatrics Society (2011) as a screening tool.
  The timed up and go combined with a cognitive task was also measured.

SECONDARY OUTCOMES:
Functional reach test | baseline
  It is a quick and simple test. It score the maximal distance one can reach forward beyond arm's length, while maintaining a fixed base of support in the standing position. The subject is asked to reach forward as far as possible without taking a step or touching the wall. It measure the ability of maintain balance during a functional task. It has been shown to be predictive of falls. It was tested with a tape measure on the wall using the head of the metacarpal of the third finger as the reference point.
Single leg stance | baseline
  This is a frequently clinical tool used to assess balance and postural steadiness. In the start position the person stand erect with arm folded across chest and the head facing straight ahead; shoes off. The subject is asked to lift one leg off the floor, based on preference of subject and keep the leg raised as long as possible without touching the other leg. Timer is stopped whether the subject's raised foot either touches the floor, makes contact with other leg or moves the stance foot to create a new base of support,if the arms move out of the test position or when a maximum balance time of 30s take place. The time was measured with a stopwatch.
Tinetti Test | baseline
  This test evaluated 13 tasks and permit the assessment of the static and dynamic balance.

OTHER OUTCOMES:
Barthel Index | baseline
  Clinical application tool of 10 items that can be administered in 2-5 minutes by a member of the medical staff or self-administered in about 10 minutes. It measure the ability to achieve certain activities without help

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain